CLINICAL TRIAL: NCT00817765
Title: Pharmacokinetic Study of Posaconazole Boosted Fosamprenavir
Acronym: EPOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Dr. D.M. Burger, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 08.03
Record Dates: First submitted 2008-12-24; First posted 2009-01-06 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: HIV Infection; Fungal Infection
Keywords: interaction; pharmacokinetics; boosting; drug-drug interaction; safety
MeSH Terms: conditions — HIV Infections; Mycoses | interventions — posaconazole; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Posaconazole alone (Active Comparator): 400mg posaconazole BID for 10 days (start on day 1 with 200mg QD, day 2 200mg BID; from day 3 onwards 400mg BID)
  Interventions: Drug: Posaconazole
- Fosamprenavir ritonavir (Active Comparator): Fosamprenavir 700mg / ritonavir 100mg BID for 10 days
  Interventions: Drug: Fosamprenavir; Drug: Ritonavir
- Fosamprenavir posaconazole (Experimental): Fosamprenavir 700mg / posaconazole 400mg BID for 10 days (start on day 1 with 200mg QD, day 2 200mg BID; from day 3 onwards 400mg BID)
  Interventions: Drug: Posaconazole; Drug: Fosamprenavir

INTERVENTIONS:
Drug: Posaconazole — Posaconazole oral solution 40mg/mL; 400mg BID treatment for 10 days, including dose escalation
  Other Names: Noxafil
  Arms: Fosamprenavir posaconazole; Posaconazole alone
Drug: Fosamprenavir — fosamprenavir tablet 700mg; 1 tablet BID for 10 days
  Other Names: Telzir / Lexiva
  Arms: Fosamprenavir posaconazole; Fosamprenavir ritonavir
Drug: Ritonavir — Ritonavir 100mg capsule; 1 capsule BID for 10 days
  Other Names: Norvir
  Arms: Fosamprenavir ritonavir

SUMMARY:
The purpose of this study is to determine the influence of posaconazole on unboosted fosamprenavir pharmacokinetics, and vice versa, in healthy volunteers.A second objective is to determine the safety of combined use of fosamprenavir with posaconazole in healthy volunteers.

DETAILED DESCRIPTION:
Infections with fungi and yeast frequently occur in patients infected with the human immunodeficiency virus type 1 (HIV-1).

Fosamprenavir is a PI that is used to treat HIV-infection in combination with ritonavir. Once hydrolyzed to amprenavir, this substance is a substrate for CYP3A4. Ritonavir is an extremely potent inhibitor of CYP3A4 and serves as a booster of the pharmacokinetics of amprenavir. Posaconazole is a very potent CYP3A4 inhibitor and therefore might enhance amprenavir pharmacokinetics in a similar way as ritonavir.

The current study is designed to test this hypothesis. When there is an indication for antifungal therapy in an HIV-infected patient, temporal replacement of ritonavir by posaconazole would be an attractive option for combined treatment of HIV and fungal infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years of age on the day of the first dosing.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to the first dose.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before the first dose) or breast-feeding female.
* Therapy with any drug (for two weeks preceding dosing), except for paracetamol.
* Subjects with an ECG with QTc interval greater than 450 ms for men, and greater than 470 ms for women at screening.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of amprenavir and posaconazole | predose and at 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours after dosing on Study Days 10, 38 and 66. Predose on study days 1, 3, 5, 8, 29, 31, 33, 36, 57, 59, 61, and 64.

SECONDARY OUTCOMES:
Adverse events (safety) due to concomitant use of fosamprenavir and posaconazole | period of interaction treatment

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Bruggemann RJ, van Luin M, Colbers EP, van den Dungen MW, Pharo C, Schouwenberg BJ, Burger DM. Effect of posaconazole on the pharmacokinetics of fosamprenavir and vice versa in healthy volunteers. J Antimicrob Chemother. 2010 Oct;65(10):2188-94. doi: 10.1093/jac/dkq280. Epub 2010 Jul 28. PMID 20667889